CLINICAL TRIAL: NCT06067568
Title: A Phase 1 Study in Healthy Subjects to Evaluate the Relative Bioavailability of Two Lutikizumab Formulations and to Evaluate Lutikizumab Pharmacokinetics, Safety, and Tolerability in Healthy Chinese Subjects
Brief Title: Relative Bioavailability of Two Lutikizumab Formulations and Pharmacokinetics, Safety, and Tolerability of Lutikizumab in Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: M24-465
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Lutikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1, Dose A (Experimental): Participants will receive a single dose of Lutikizumab Dose A.
  Interventions: Drug: Lutikizumab Dose A
- Part 1, Dose B (Experimental): Participants will receive a single dose of Lutikizumab Dose B.
  Interventions: Drug: Lutikizumab Dose B
- Part 2 (Experimental): Han Chinese participants will receive a single dose of Lutikizumab.
  Interventions: Drug: Lutikizumab Dose A

INTERVENTIONS:
Drug: Lutikizumab Dose A — Injection; subcutaneous (SC)
  Arms: Part 1, Dose A; Part 2
Drug: Lutikizumab Dose B — Injection; subcutaneous (SC)
  Arms: Part 1, Dose B

SUMMARY:
The purpose of this study is to compare the bioavailability of two different formulations of lutikizumab, and to assess adverse events (AEs) and how lutikizumab moves through the body in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers aged between 18 and 60 years.

  -- Part 2 only: Participant must be first-generation Han Chinese of full Chinese parentage residing outside of China. Participant must maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.
* BMI <= 18.0 to <= 29.9 kg/m^2 after rounding to the tenths decimal, at screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Use any medications, vitamins, and/or herbal supplements within the 2 week period or 5 half-lives (whichever is longer) prior to study drug administration.
* History of: epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic ,gastrointestinal, hematologic, demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease, glaucoma, psychiatric disease or disorder, or any uncontrolled medical illness.
* Prior exposure to lutikizumab.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Lutikizumab | Up to Day 8
  Cmax of lutikizumab will be assessed.
Time to Cmax (Tmax) of Lutikizumab | Up to Day 8
  Tmax of lutikizumab will be assessed.
Apparent Terminal Phase Elimination Rate Constant (β) of Lutikizumab | Up to Day 8
  Apparent terminal phase elimination rate constant (β) of lutikizumab will be assessed.
Terminal Phase Elimination Half-life (t1/2) of Lutikizumab | Up to Day 8
  Terminal phase elimination half-life (t1/2) of lutikizumab will be assessed.
Area under the Serum Concentration-time Curve (AUC) from Time 0 to the Time of the Last Measurable Concentration (AUC0-t) of Lutikizumab | Up to Day 8
  AUC0-t of lutikizumab will be assessed.
AUC from Time 0 to Infinity (AUC0-inf) of Lutikizumab | Up to Day 8
  AUC0-inf of lutikizumab will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 71
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Altasciences Clinical Los Angeles, Inc /ID# 260986, Cypress, California
  - Acpru /Id# 259029, Grayslake, Illinois
  - PPD Clinical Research Unit - Austin /ID# 260141, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-465